CLINICAL TRIAL: NCT01857180
Title: Introduction of a Comprehensive Training Curriculum in Laparoscopic Surgery for Medical Students: a Randomized Trial.
Brief Title: Comprehensive Laparoscopic Curriculum for Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Med Student Lap Curriculum
Record Dates: First submitted 2013-05-15; First posted 2013-05-20 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Education; Laparoscopic Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curriculum (Experimental): Participants in the curriculum group took part in a structured, comprehensive curriculum consisting of a 1 hour didactic cognitive component, a 1 hour didactic non-technical (team-based skills) component, and 6 hours of structured technical skills practice in peg transfer, intracorporeal suture, and VR simulator tasks. Participants had the opportunity to ask questions and engage in discussion with experts after the didactic sessions, and received subjective feedback from circulating residents in addition to objective feedback in the technical skills tasks.
  Interventions: Other: Curriculum
- Self-directed (No Intervention): Participants in the control (self-directed) group took part in 8 hours of self-directed learning with written materials for cognitive and non-technical skills components and unstructured surgical simulation practice of technical skills with only objective feedback from the simulator for the VR tasks or time for the peg transfer and intracorporeal suture tasks.

INTERVENTIONS:
Other: Curriculum
  Arms: Curriculum

SUMMARY:
Laparoscopic surgery has become the standard approach to a vast variety of surgical procedures. Due factors such as 2D- to 3D conversion, reduced tactile sensation, amplification of tremor and fulcrum effect of the abdominal wall, surgeons require a different set of skills than in open access surgery. Acknowledging this, several comprehensive curricula have been developed to teach basic skills as well as advanced laparoscopic procedures. Despite a recent emphasis on early exposure of medical students to surgery no designated curricula have been developed to introduce medical students to the technique of laparoscopic surgery.

Participation in an introductory curriculum in laparoscopic surgery results in improved cognitive and technical performance compared to self-directed learning. The greater homogeneity and fewer dropouts amongst those in the curriculum group suggest that a structured curriculum is essential in ensuring standardization of clinically relevant training. An introductory curriculum for medical students should be delivered in a structured and standardized fashion prior to clinical exposure in order to maintain motivation and enhance learning.

ELIGIBILITY:
Inclusion Criteria:

* first and second year medical students

Exclusion Criteria:

* previous exposure to laparoscopy or laparoscopic simulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Cognitive Knowledge | 1 week
  Participants' basic laparoscopic knowledge was assessed regarding topics such as advantages and disadvantages, patient selection considerations, equipment, anesthesia, patient positioning, pneumoperitoneum, and post-op care. Assessment was by a multiple choice test.
Team-based (non-technical) skills | 1 week
  Participants' attitudes towards team based skills, namely team structure, leadership, situational awareness, and communication were assessed by the Team-STEPPS Teamwork Attitudes Questionnaire (T-TAQ).
Technical Skills | 5 weeks
  Participants' technical skills were assessed as they performed peg transfer, intracorporeal suture, and virtual reality simulator tasks (grasping, cutting, and clipping). Peg transfer and intracorporeal suture were assessed by time and errors, while VR tasks were assessed by the simulator's pre-set metrics.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Toronto, Toronto, Ontario, Canada